CLINICAL TRIAL: NCT06346522
Title: Efficacy of Gabapentin Versus Trospium Chloride for Prevention of Catheter-related Bladder Discomfort (CRBD) Inside the Intensive Care Unit (ICU): a Prospective, Randomized,Comparative Clinical Study
Brief Title: Gabapentin Versus Trospium Chloride for Prevention of a Catheter-related Bladder Discomfort Inside the ICU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU R37/2024
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2024-03

CONDITIONS: Catheter-related Bladder Discomfort (CRBD)
Keywords: Catheter-related bladder discomfort (CRBD); Gabapentin; Trospium chloride; Intensive Care Unit (ICU); Postoperative care
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, comparative, clinical trial study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- -Group G (40 patients): Gabapentin (Active Comparator): After the patient will regain feeding, the patients will take with sips of water Gabapentin (Gaptin ®) 400mg oral capsule once in the first 24 hour after icu admission
  Interventions: Drug: Gabapentin (Gaptin ®) 400mg oral capsule once
- -Group T (40 patients): Trospium chloride slow release (Active Comparator): After the patient will regain feeding, the patients will take with sips of water Trospium chloride slow release (Trospikan ® SR) 60mg oral capsule once in the first 24 hour after icu admission
  Interventions: Drug: Trospium chloride slow release (Trospikan ® SR) 60mg oral capsule
- Group C (40 patients): Non-pharmacological standard of care control group (No Intervention): Non-pharmacological standard of care control group who administered nothing

INTERVENTIONS:
Drug: Gabapentin (Gaptin ®) 400mg oral capsule once — After the patient will regain feeding, the patients will take with sips of water Gabapentin (Gaptin ®) 400mg oral capsule once in the first 24 hour after icu admission
  Other Names: Gaptin ®
  Arms: -Group G (40 patients): Gabapentin
Drug: Trospium chloride slow release (Trospikan ® SR) 60mg oral capsule — After the patient will regain feeding, the patients will take with sips of water Trospium chloride slow release (Trospikan ® SR) 60mg oral capsule once in the first 24 hour after icu admission
  Other Names: Trospikan ® SR
  Arms: -Group T (40 patients): Trospium chloride slow release

SUMMARY:
Catheter-related bladder discomfort (CRBD) is a frequent complaint after urinary bladder catheterization which is commonly done in the perioperative period. CRBD shows similar symptoms to overactive bladder (OAB); so, drugs used for the management of OAB could influence symptoms of CRBD. Trospium chloride and gabapentin are effective in managing patient with OAB even the resistant cases. We will evaluate and compare the efficacy of both oral trospium and gabapentin on prevention of CRBD in the postoperative period in the ICU in in patients undergoing spinal surgery and requiring intraoperative catheterization of the urinary bladder.

DETAILED DESCRIPTION:
* Study will be conducted in the intensive care units (ICU) of Ain Shams University Hospitals, Cairo, Egypt
* After satisfactory pain control and full recovery in the postanesthesia care unit (PACU), the patient will be transferred to the ICU as a case of postoperative care after elective spinal diskectomy surgeries (cervical, dorsal or lumber) with removal of the damaged portion of the herniated or degenerated disks. Admission to ICU will be for medical, surgical or anesthesia related causes.
* Standard monitoring devices via GE monitor will be connected to the patient as electrocardiogram (ECG) for heart rate (beats/min), pulse oximetry for (SPO2 as a percentage) and non-invasive blood pressure (NIBP) (mmHg).Temperature of the patient in Celsius (◦C), random blood sugar (mg/dl) and urine output (ml/hour) will be monitored also. Follow-up by standard postoperative laboratory tests will be done too.
* After the patient will regain feeding according to the European Society for Clinical Nutrition and Metabolism (ESPEN) guidelines [1],the consented and enrolled 120 patients will be randomly assigned to one of the following groups and oral drug will be taken with sips of water:
* Group G (40 patients): Gabapentin (GaptinR) 400mg oral capsule
* Group T (40 patients): Trospium chloride slow release (TrospikanR SR) 60mg oral capsule
* Group C (40 patients): Non-pharmacological standard of care control group who administered nothing
* Incidence and severity of CRBD will be assessed by 4-point severity scale developed by Agarwal in1,2,6,12,24 hours after the study drugs intake . Assessment of pain severity and control will be done by using Numerical Pain Rating Scale (NPRS) and measuring total fentanyl requirements in the 1st 24h in micrograms (µg/day). Side effects of the study drugs will be recorded and managed accordingly with the use of Ramsay sedation score to assess sedation level one hour after the study drugs intake .
* Patients will continue their monitored care in the ICU till the control of the causes of their ICU admission or their end.
* Demographic data, causes for postoperative care in the ICU (Medical, surgical or anesthesia related) and spine surgery site and number for each (cervical, dorsal, lumber) will be collected and recorded.The collected study data results will be revised, electronically recorded in datasheet, coded, tabulated, analyzed, and processed using the proper computerized statistical package program. Suitable statistical analysis will be done according to the type of data obtained for each parameter with comparison between groups to identify any significant differences between them

ELIGIBILITY:
Inclusion Criteria:

* Both males and females with age 20-65 years
* American Society of Anesthesiologists (ASA) physical status class I, II or III.
* Patients will undergoing elective spinal surgery and will require catheterization of the urinary bladder.

Exclusion Criteria:

* known allergy to the study drugs or patient refusal.
* Urinary bladder pathology as overactive bladder (frequency more than 3 times in the night or more than 8 times in 24 h), bladder outflow obstruction, urinary tract infection or malignancy
* Preoperative neurological bladder and/or bowel involvement secondary to spinal cord compression.
* Chronic opioids use for chronic pain, drugs or alcohol abuse
* Moderate to severe hepatic disease, renal impairment with creatinine clearance (CrCl) less than 30 ml/minute
* Narrow angle glaucoma
* Psychiatric diseases
* Gastrointestinal obstructive conditions as severe chronic constipation or ileus

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
The incidence (yes/no) and severity of catheter-related bladder discomfort (CRBD) in 1,2,6,12,24 hours after the study drugs intake | First 24 hours after the study drugs intake
  Severity of CRBD will be assessed and recorded by a CRBD 4-point severity scale developed by Agarwal et al as following:
  1. No discomfort
  2. Mild: urinary urgency or suprapubic discomfort reported by the patient on questioning only
  3. Moderate: urinary urgency or suprapubic discomfort reported by the patient themselves without being questioned and not accompanied by behavioral changes
  4. Severe: urinary urgency or suprapubic discomfort reported by the patient themselves and accompanied by behavioral changes such as attempts to remove the catheter, verbal responses, and restless movements of extremities) [2]

SECONDARY OUTCOMES:
Total fentanyl requirements in micrograms (µg) | First 24 hours after the study drugs intake
  Total fentanyl requirements in the 1st 24h after study drugs intake in micrograms (µg/day)
Numerical Pain Rating Scale (NPRS) (0-10) | First 24 hours after the study drugs intake
  NPRS for measurement of surgical pain intensity. It consists of a 10 cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').NPRS will be assessed at 1,2,6,12,24 hours after the study drugs intake.
Side effects of the study drugs | First 24 hours after the study drugs intake
  They includes:
  * Nausea and vomiting
  * Dry mouth
  * Light headedness or confusion
  * Headache
  * Tachycardia
  * Blurred vision
  * Facial flushing
  * Agitation
  * Constipation
Ramsay sedation score | After one hour of the study drugs intake
  Ramsay sedation score [3].It will be assessed after one hour of the study drugs intake
  Score Sedation level
  1. Awake; agitated or restless or both
  2. Awake; cooperative, oriented, and tranquil
  3. Awake but responds to commands only
  4. Asleep; brisk response to light glabellar tap or loud auditory stimulus
  5. Asleep; sluggish response to light glabellar tap or loud auditory stimulus
  6. Asleep; no response to glabellar tap or loud auditory stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Mohamed, MD, Principal Investigator — Ain Shames University
Locations (1):
- Ain Shams University-Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and analyzed during the current study are available from the corresponding author on reasonable request, with hiding of identities of participants or any personal information.

REFERENCES:
- [Background] Weimann A, Braga M, Carli F, Higashiguchi T, Hubner M, Klek S, Laviano A, Ljungqvist O, Lobo DN, Martindale RG, Waitzberg D, Bischoff SC, Singer P. ESPEN practical guideline: Clinical nutrition in surgery. Clin Nutr. 2021 Jul;40(7):4745-4761. doi: 10.1016/j.clnu.2021.03.031. Epub 2021 Apr 19. PMID 34242915
- [Background] Agarwal A, Dhiraaj S, Singhal V, Kapoor R, Tandon M. Comparison of efficacy of oxybutynin and tolterodine for prevention of catheter related bladder discomfort: a prospective, randomized, placebo-controlled, double-blind study. Br J Anaesth. 2006 Mar;96(3):377-80. doi: 10.1093/bja/ael003. Epub 2006 Jan 16. PMID 16415311
- [Background] Ramsay MA, Savege TM, Simpson BR, Goodwin R. Controlled sedation with alphaxalone-alphadolone. Br Med J. 1974 Jun 22;2(5920):656-9. doi: 10.1136/bmj.2.5920.656. PMID 4835444